CLINICAL TRIAL: NCT04200859
Title: The Effect of Different Cold Application Materials on Pain During Chest Tube Removal: A Randomized Controlled Trial
Brief Title: Effect of Cold Application Materials on Pain During Chest Tube Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gulay ALTUN UGRAS, Associate Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mersin University
Record Dates: First submitted 2019-12-10; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Local Application / Packing Too Cold
Keywords: chest tube,; chest tube removal; pain; cold aplication; nursing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Prospective, parallel three armed, randomized controlled trial
Masking Description: No blinding in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cold application with ice pack (Experimental): Before the chest tube was removed, two ice packs with a size of 15.5x9cm were inserted around the chest tube so as to make as much contact as possible
  Interventions: Other: Cold application
- Cold application with gel pad group (Experimental): Before the chest tube was removed, a gel pad with a radius of 15 cm was completely inserted around the chest tube
  Interventions: Other: Cold application
- Control group (No Intervention): Routine analgesic drugs are not administered to patients before removal of the chest tube in thoracic surgery clinic. However, analgesic is performed according to the severity of pain after the procedure.

INTERVENTIONS:
Other: Cold application — cold application using ice pack/gel pad in the control of pain experienced during chest tube removal
  Arms: Cold application with gel pad group; Cold application with ice pack

SUMMARY:
Background: Despite being an important treatment intervention, chest tube causes severe pain during removal because it attaches to the endothelium in the chest cavity.

Objectives: This study aimed to determine the effectiveness of cold application with ice pack and gel pad in the control of pain experienced during chest tube removal.

Design: Prospective, parallel three armed, randomized controlled trial. Settings: The study was conducted in athoracic surgery unit of a university hospital.

Methods: The sample of this study consisted of 180 patients in two experimental groups and one control group.The patients were randomly assigned by a computer program to either intervention groups (ice pack or gel pad) or control group.One experimental group received cold application using ice pack and the other received cold application using gel pad until the skin temperature of all the patients fell to 13.6°C. The control group did not receive any intervention. Pain severity was assessed with Numerical Rating Scale (NRS) before chest tube removal, at the end of the procedure and 15 minutes after the procedure. Data was analyzed using descriptive statistics, chi-square, student t-test in independent groups, one-way analysis of variance (ANOVA), and repeated measures ANOVA.

DETAILED DESCRIPTION:
This study was aimed to determine which cold application material is more effective in pain control of patients during chest tube removal process.

The primary outcomes measures of this study were the effect of cold application materials on severity of pain.The secondary outcome measures of this study were duration of cold application and analgesic requirements of the patients.

Procedure Before removal of chest tube, nurse researcher (DS) who is working in the thoracic surgery clinic as a nurse, explained aim of study and take informed consent all patients. Data were collected with Patient Information Form and NRS.

Patient Information Form was filled out for each using the information obtained from patients/patients' relatives, patient files and health professionals of the clinic and the patients' pain severity was measured with NRS.

The patients were randomly assigned by a computer program to either intervention groups (ice pack or gel pad) or control group. Before the chest tube was removed, nurse researcher (DS) made cold application with ice pack the first experimental group and cold application with gel pad the second experimental group. The control group did not receive any intervention. Since the cold application temperature should be reduced to 13.6 °C in order to have local analgesic effect in both of the experimental groups the patient's skin temperature was measured at one-minute intervals by using an infrared non-contact thermometer (Microlife Non-Contact, Switzerland) with a wide measurement range (0-100 °C) and a measurement time of three seconds. This application was terminated when the temperature was 13.6 °C and the chest tube was removed by the physician.

Pain severity of all the patients was measured with NRS immediately after and 15 minutes after chest tube removal.

ELIGIBILITY:
Inclusion Criteria:

* had chest tube
* Must be conscious, orientated and cooperated
* Must be able to speak and understand Turkish

Exclusion Criteria:

* Psychiatric disease
* Language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
effect of cold application materials on severity of pain | Change from first NRS at 15 minutes
  Numerical Rating Scale: The scale was used to determine the severity of pain during chest tube removal process. On this scale, patients are asked to describe their pain with numbers, with "0" indicating "no pain" and "10" indicating "the worst, unbearable pain"

SECONDARY OUTCOMES:
effect of cold application materials on duration of cold application | 30 minutes
  The Patients Information Form was used to determine patients duration of cold application. How many minutes of cold application material applied
effect of cold application materials on analgesic requirements of the patients | up to 6 hours
  The Patients Information Form was used to determine presence of analgesic administration after chest tube removal, time passed between the last analgesic time and chest tube removal time and time passed between chest tube removal time and the first analgesic administration time.

IPD SHARING:
Plan to Share IPD: Undecided